CLINICAL TRIAL: NCT05393765
Title: The Evaluation of the Effect of an Interactive Web-based Program That Supports Nurse-led Self-regulation in the Management of Multiple Sclerosis
Brief Title: The Effect of an Interactive Web-based Program in the Management of Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Ayyuce Tuba Kocak, Research assistant, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/33
Record Dates: First submitted 2022-05-20; First posted 2022-05-26 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Self-Management; Nursing; Self-Regulation
MeSH Terms: conditions — Multiple Sclerosis; Self-Control

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial with a two-group pre-test and post-test design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): Experimental: Intervention group "Yönetebilirim" Before the initiation of the program, patients who visit the outpatient clinic will be evaluated according to the inclusion-exclusion criteria, their consent will be obtained, and pre-tests will be administered. Then, randomization will be performed and participants will be assigned to the experimental and control groups. Participants in the experimental group will be registered on the web-based program. The individuals in the experimental group will use "Yönetebilirim" for 8 weeks as of the time the program is put into use. "Yönetebilirim" consists of modules and consultancy services. Participants will be able to watch informative videos as much as they want for 8 weeks and receive consultancy service if they wish.
  Interventions: Behavioral: Yönetebilirim
- Control (No Intervention): The control group will receive standard care without any intervention. The group will not receive any other intervention.

INTERVENTIONS:
Behavioral: Yönetebilirim — "Yönetebilirim" is an interactive web-based program developed to improve the self-management skills of individuals with MS by supporting self-regulation under the leadership of nurses.
  Arms: experimental

SUMMARY:
This study aimed to investigate the effect of an interactive web-based program that supports nurse-led self-regulation in the management of Multiple Sclerosis (MS) on the self-management, fatigue and anxiety levels of patients with Multiple Sclerosis.

DETAILED DESCRIPTION:
Detailed Description: Individuals with Multiple Sclerosis are diagnosed at a young age and face a long-term, heterogeneous disease process with effects on multiple functional areas. As in other chronic diseases, individuals with MS need to develop self-management skills in order to be integrated into society, to have an increased quality of life, to reduce the burden of symptoms, to prevent disability, and to maintain psychosocial well-being. In order to improve self-management skills, it is important for the healthcare team to have a supervisory and educational role and to carry out the clinical and social follow-up of these individuals closely. Studies have shown that those with MS do not generally use health services except for the attack periods or they have problems in reaching the health care team due to reasons such as fatigue and disability. It is reported that individuals with MS mostly seek information on the Internet, on social media or from peers, and they do not consult the healthcare team about this inaccurate or insufficient information. All these factors clearly indicate that digital health (e-health) services should become widespread alongside traditional health services in order to improve the self-management skills of individuals with MS.

It is seen in the literature that various web-based programs with different interfaces and features have been developed by different healthcare team members for individuals with MS; however, many of these programs have not been evaluated in randomized controlled studies and are not nurse-led. MS is considered as a very long journey for individuals and their families, and nurses accompany individuals with MS and their families as a leading force to support self-management throughout this journey. No interactive web-based programs have been developed to support the self-management skills of individuals with MS in Turkey. Considering that this is an important gap, an interactive web-based program named "Yönetebilirim", which supports self-regulation under the leadership of nurses, was developed. This study aims to evaluate the effect of "Yönetebilirim" on self-management, fatigue and anxiety levels of individuals with MS with a randomized controlled design.

Yönetebilirim "Yönetebilirim" is an interactive web-based program developed to improve the self-management skills of individuals with MS by supporting self-regulation under the leadership of nurses. The program was shaped in accordance with action research in a collaborative design and was implemented between February 2021 and May 2022 with the approval of the non-interventional clinical research ethics committee of a university (2021/61). Under the coordination of the action researcher (program coordinator), the components of the web-based program were shaped by individuals with MS, nurses caring for individuals with MS, and software specialists. The self-regulation strategies formed the theoretical basis of the web-based program. The domain name of the program has been taken and its address has been determined as "yonetebilirim.com".

The program consists of modules and consultancy services. Modules There are a total of 10 modules in the program and the modules are presented under two headings as "Informative" and "Interactive". The topics of the modules are as follows: Recognizing MS and Attack management, Coping with fatigue, Sexual health, Bladder and Urinary problems, Self-monitoring, Healthy lifestyle behaviors, Importance of physiotherapy, MS Stories and Laughter therapy. The speakers in the modules are a specialist neurologist, academician nurses, specialist nurses, a specialist physiotherapist, and a laughter therapist who voluntarily agreed to support the program. The modules consist of discussion sessions based on the program coordinator's questions and the speakers' answers. The content of the videos was created by the speakers according to their fields of expertise. The informative modules include video recordings and written documents aiming at sharing information. The interactive modules consist of interactive live webinars created to increase motivation.

Consultancy Services After the participants are accepted to the program, they will be able to access the program with their own username and password. Participants will be able to receive counseling from the nurse with a written message using the "Consult" link on the main screen of the program, and the nurse will be able to answer questions through the system. If they wish, participants will be able to make an appointment to meet online with the video conference method by clicking on the "Request a Meeting" link.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed with Multiple Sclerosis,
* Expanded Disability Status Scale (EDSS) score below 5,
* Be in the 7-12 age range18-65,
* Having the ability to read and write,
* To be able to communicate in Turkish
* Being able to access and use the Internet (computer, tablet, mobile phone)

Exclusion Criteria:

* To have received steroid treatment for an attack in the last month
* Having a psychiatric diagnosis (schizophrenia, bipolar affective disorder etc.)
* Having advanced cognitive problems
* Being visually and hearing impaired.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Change in self-management | Baseline and 8 weeks after patient inclusion
  The Multiple Sclerosis Self-Management Scale (MSSM) will be used to assess self-management knowledge and behavior of individuals with MS comprehensively and psychometrically. The MSSM consists of 24 Likert-type items with re-sponses as follows: disagree completely (1 point), somewhat disagree (2 points), neither agree nor dis-agree (3 points), somewhat agree (4 points), and agreecompletely (5 points). The MSSM includes 5 subscales: healthcare providerrelationship/communication, treatment adherence/barriers, social/family support, MS knowledge and information, and health maintenance behavior. Total score ranges between 0 and 100, and a higherscore indicates a higher degree of self-management.

SECONDARY OUTCOMES:
Fatigue Severity Scale | Baseline and 8 weeks after patient inclusion
  The scale, which evaluates fatigue in the last month, consists of 9 items and is a 7-point Likert type. The scale has only one sub-dimension and each question is evaluated between 1-7 points. The lowest score that can be obtained from the salep item is 1 and the highest score is 7. The total score in the scale is calculated by taking the average of 9 items. A score of four or more generally indicates severe fatigue. As the score obtained from the scale increases, the degree of fatigue also increases.
State-Trait Anxiety Inventory (STAI) | Baseline and 8 weeks after patient inclusion
  State-Trait Anxiety Inventory (STAI) is self-report questionnaire consists of two subscales each containing 40 items, 20 item state, 20 item trait. All items are rated on a 4-point scale. Higher scores indicate greater anxiety. The scale is evaluated over the total score, and as the score obtained from the scale increases, the level of anxiety also increases. In the score calculation, the score obtained for the direct statements is subtracted from the score obtained for the reverse statements. This value is added to the constant value of 35 for the Trait Anxiety Scale. Bigger score indicates high anxiety level; small score indicates low anxiety level.
System Usability Scale | 8 weeks after patient inclusion
  System Usability Scale consists of a 10 item questionnaire with five response options for respondents; from Strongly agree (5 point) to Strongly disagree (1 point). For each of the odd numbered questions, subtract 1 from the score. For each of the even numbered questions, subtract their value from 5.Take these new values which you have found, and add up the total score. Then multiply this by 2.5. The scores of scale are 0-100. The scale score above a 68 would be considered above average and anything below 68 is below average.
Program Usage Level Tracking Form | 8 weeks after patient inclusion
  In the research, the level of use of "Yönetebilirim" and the participation status of the participants in the experimental group will be evaluated with a 7-question program usage level follow-up form created by the researcher. The form will be filled by the researcher according to the data recorded by the program.

CONTACTS AND LOCATIONS:
Overall Officials: Selda Arslan, Phd, Study Director — Necmettin Erbakan University Faculty of Nursing; Ayyüce Tuba Koçak, MSC, Principal Investigator — Selcuk University Faculty of Nursing
Locations (1):
- Selcuk University, Selçuklu, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 3 mounts later